CLINICAL TRIAL: NCT04910126
Title: Doxorubicin（A）Plus Camrelizumab(C) Versus Doxorubicin Alone for the First-line Treatment(T) of Select Type of Adcanced Soft Tissue Sarcoma(ACTS): a Randomised Controlled Multi Centers Trial
Brief Title: Camrelizumab Plus Doxorubicin for the First Line Treatment of Adcanced Soft Tissue Sarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Jing Chen, Director, Head of Sarcoma Department , Principal Investigator, Clinical Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTS
Record Dates: First submitted 2021-05-24; First posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Soft Tissue Sarcoma; Neoplasms, Connective and Soft Tissue; Sarcoma Metastatic; Sarcoma,Soft Tissue
MeSH Terms: conditions — Sarcoma; Neoplasms, Connective and Soft Tissue | interventions — camrelizumab; Doxorubicin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experiment group (Experimental): adriamycin and Camrelizumab
  Interventions: Drug: Camrelizumab; Drug: Adriamycin
- control group (Active Comparator): adriamycin
  Interventions: Drug: Adriamycin

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab 200mg q3w up to 2 years
  Other Names: C
  Arms: experiment group
Drug: Adriamycin — adriamycin 20mg/m2 d1-3 q3w maximum 6 cycles
  Other Names: A

SUMMARY:
To evaluate the efficacy and safety of the combination of adriamycin and Camrelizumab in the first-line treatment of advanced soft tissue sarcoma

ELIGIBILITY:
Inclusion Criteria:

- 1) Patients with advanced soft tissue sarcoma (pathologically confirmed undifferentiated pleomorphic sarcoma/synovial sarcoma/leiomyosarcoma/liposarcoma) not suitable for surgery; 2) Aged ≥ 18 years old, < 60 years old; 3) Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1, amputees can be 0-2; 4) Expected survival > 6 months; 5) Adequate organ and bone marrow function, defined as follows: ① Blood routine (14 days before screening without blood transfusion, without G-CSF, without drug correction): neutrophil count (ANC) ≥ 1.5 × 10^9/L; platelet count (PLT) ≥ 100 × 10^9/L; hemoglobin (Hb) ≥ 100 g/L; ② Blood biochemistry: serum creatinine (Cr) ≤ 1.5 × upper limit of normal (ULN) or creatinine clearance ≥ 60ml/min; total bilirubin (TBIL) ≤ 1.5 × ULN; aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level ≤ 2.5 × ULN, The subjects with liver metastasis should be ≤ 5 × ULN; ③ Coagulation function: international normalized ratio (INR) ≤ 1.5, prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN; ④ Urinalysis: urine protein < 2 +; if urine protein ≥ 2 +, the 24-hour urine protein quantification must be ≤ 1g; ⑤ thyroid stimulating hormone (TSH) ≤ ULN and ≥ LLN; if abnormal, T3 and T4 levels should be investigated, normal T3 and T4 levels can be included.

6) ECG is basically normal, no myocardial ischemia performance, no history of arrhythmia requiring drug intervention, echocardiography LVEF ≥ 50%; 7) no autoimmune diseases; 8) can provide tissue samples for biological testing; 9) have measurable lesions according to RECIST1.1 criteria; 10）Agree and have signed informed consent, willing and able to comply with scheduled visits, study treatment, laboratory tests and other test procedures.^

Exclusion Criteria:

* 1) Patients who have previously received anthracycline treatment; 2) Patients who have previously received immunotherapy such as anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA4, etc.; 3) Patients who are known to be allergic to recombinant humanized anti-PD-1 monoclonal antibody drugs and their components; 4) Patients with New York Heart Association (NYHA) score of more than II heart disease (including grade II); 5) Patients with mental or neurological disorders or do not cooperate; 6) Patients who have received other anti-tumor therapy 4 weeks before enrollment, including but not limited to surgery, radiotherapy, chemotherapy, targeted therapy, immunotherapy, etc.; 7) Patients who have used immunosuppressive drugs within 14 days before enrollment. Does not include nasal spray and inhaled corticosteroids or physiological doses of systemic steroids (i.e., no more than 10 mg/day prednisolone or other corticosteroids at physiological doses of the same drug); 8) any active autoimmune disease or history of autoimmune disease (subjects with vitiligo or asthma that has been completely relieved in childhood and currently does not require medical intervention can be included), or known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.

  9) Known allergy to the study drug or any of its excipients; or severe allergic reactions to other monoclonal antibodies; 10) Patients with central nervous system metastasis; 11) Patients with severe systemic infection (who need intravenous antibiotics, antifungal or antiviral drugs) within 4 weeks before enrollment, or body temperature ≥ 38.0℃; 12) Patients received live vaccination within 4 weeks before the start of treatment; 13) HIV infection, HCV antibody positive and HCV RNA higher than the lower limit of detection of the analytical method, HBsAg or HBcAb positive and HBV DNA positive (quantitative detection limit of 500 IU/ml); 14) History of active pulmonary tuberculosis; 15) Patients who had been diagnosed with any other malignant tumor within 3 years before enrollment, except for adequately treated basal cell or squamous cell skin cancer or cervical carcinoma in situ; 16) Pregnant women or lactating women, or patients who plan to become pregnant during the study period or within one year after the use of the study drug; 17) Patients who participating in the trial is not in their best interest (such as endangering their health) or will hinder the evaluation of the trial protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2020-11-12 (Actual); Primary Completion 2023-01-12 (Estimated); Study Completion 2023-11-12 (Estimated)

PRIMARY OUTCOMES:
PFS | up to three years
  progression-free survival

SECONDARY OUTCOMES:
OS | up to three years
  overall survival
ORR Objective Response Rate（ORR） | up to one year
  Objective Response Rate
DOR | up to two years
  Duration of Response
AE | up to three years
  treatment related adverse events, TRAEs

CONTACTS AND LOCATIONS:
Overall Officials: Jing Chen, MD, PhD, Study Chair — Huazhong University of Science and Technology
Locations (1):
- Union Hospital，Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No